CLINICAL TRIAL: NCT06866847
Title: Muscle Strength, Muscle Endurance, Lower Extremity Function, Aerobic Capacity, Pressure Pain Threshold and Edema in Women with Lipedema: a Case-Control Study
Brief Title: Muscle Strength, Muscle Endurance, Lower Extremity Function, Aerobic Capacity, Pressure Pain Threshold and Edema in Women with Lipedema
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ilke Keser, Prof. Dr., Gazi University
Other Study IDs: Lipedema/Haspolat M
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Lipedema; Healthy
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- study group: Women diagnosed with lipedema
- control group: Women over the age of 18 who do not have any cardiovascular, orthopedic and/or neurological problems that may affect physical capacity and who do not have diseases such as heart failure or renal failure that may cause general or localized edema.

SUMMARY:
Lipedema is a chronic progressive disease that causes disproportionate, painful extremities with abnormal fat distribution. Lipedema is known to cause physical and psychosocial disorders in individuals, but there are very limited studies on this subject. The aim of this study is to evaluate muscle strength, muscle endurance, lower extremity function, aerobic capacity, pressure pain threshold and edema parameters in individuals diagnosed with lipedema and to compare them with individuals without lipedema. Volunteer women aged 18 years and older with lipedema (study group) and without lipedema (control group) will be included in the study. After recording the demographic information of the patients, lower extremity muscle strength will be assessed with the K-force handheld dynamometer, lower extremity muscle endurance with the 30 Second Sit-to-Stand Test, lower extremity function with the Lower Extremity Functional Scale, aerobic capacity with the 6-Minute Walking Test, pressure pain threshold with the Baseline algometer, and edema with the moisturemeter. Data from the study and control groups will be recorded in the SPSS program and compared using the appropriate statistical method.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 diagnosed with lipedema

Exclusion Criteria:

* Having cardiovascular, orthopedic and/or neurological problems that may affect physical capacity

  * Having diseases such as heart failure, kidney failure that may cause general or localized edema

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with lipedema in Ankara/TURKEY
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of Muscle Strength | only one time
  The individuals' gluteus maximus, hip flexor, abductor and knee extensor strength in their dominant extremities will be assessed with a K-force handheld dynamometer (Montpellier, France). In the assessment, the individual will be positioned in a prone position for the gluteus maximus muscle test, in a sitting position for the hip flexor and extensor muscles test and in a side-lying position for the hip abductors test, and the dynamometer will be stabilized as specified in the K-Force manual, and the individual will be asked to apply maximum effort against the dynamometer. The measurements will be repeated 3 times and the maximum value will be recorded in kg.
Assessment of Lower Extremity Muscle Endurance | only one time
  Lower extremity muscle endurance will be assessed with the 30-Second Sit-Stand Test. In this test, the individual will sit on a chair with their back supported. The individual will then be asked to stand up and sit down again with their back straight for 30 seconds, and the number of times this cycle is repeated within 30 seconds will be recorded.
Assessment of Lower Extremity Function | only one time
  It will be evaluated with the Lower Extremity Functional Scale. The Lower Extremity Functional Scale is a questionnaire developed to evaluate individuals' lower extremity functions, abilities and activity limitations. Scoring is between 0-80. Higher scores indicate better function. It is based on the individual's self-assessment and personal statement. The Turkish version of the scale was developed by Çankaya et al. and reported to be valid and reliable.
Assessment of Aerobic Capacity | only one time
  It will be evaluated with the 6 Minute Walking Test. During this test, the individual is asked to walk as fast as he can in a 30-meter corridor for 6 minutes and the total walking distance is recorded in meters.
Assessment of Pressure Pain Threshold | only one time
  A digital algometer (Baseline) will be used to assess the pain threshold. The algometer will be calibrated before the assessment. A 1 cm2 probe will be used for the measurements. The midpoint of the quadriceps and tibia will be marked before the measurement. The measurement will be repeated 3 times at 5-second intervals and the average value will be recorded. The algometer will be placed at a right angle to each point, participants will be asked to report the presence of pain by saying "yes" and the value on the device will be recorded as the pain threshold when they first feel pain at the point of touch. There will be a 5-second interval between measurements
Assessment of Edema | only one time
  Local tissue water percentage of individuals will be measured with the Moisturemeter-d compact (MMDc, Delfin Technologies, Kuopio, Finland) device. This device calculates the percentage of water under the skin by touching the reference points from the skin surface. The reference points were determined as the medial of 35 cm above the heel (calf) on both legs, the medial of 3 cm proximal to the patella (medial knee) and the lateral of 20 cm above the line drawn from 3 cm proximal to the patella to the SIAS (lateral hip) (6). 3 measurements will be made for each reference point and the average of these measurements will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Health Sciences, Ankara, Turkey (Türkiye)